CLINICAL TRIAL: NCT03534375
Title: Gender Differences in Risk-proneness, Gratification Delay, Self-control, Self-efficacy, Executive Functions and Their Neurophysiological and Neuroanatomical Correlates in Early Adolescents
Brief Title: Gender Differences of Neuroanatomical and Neurophysiological Correlates of Risk-proneness in Early Adolescents
Status: Completed | Type: Observational
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB2017-914
Record Dates: First submitted 2018-05-09; First posted 2018-05-23 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Gender; Early Adolescent Behavior
MeSH Terms: conditions — Coitus; Adolescent Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female Early Adolescents
  Interventions: Other: The study is an observational cross sectional study
- Male Early Adolescents
  Interventions: Other: The study is an observational cross sectional study

INTERVENTIONS:
Other: The study is an observational cross sectional study — An intervention will not be performed

SUMMARY:
Risk-taking in early adolescence have has been found to be normative and even formative as it might fulfill the youth's needs to experiment different sensations, make independent decisions and learn from their consequences. Several theoretical models have suggested that male and female adolescents differ in risk-taking as a product of individual/contextual factors and neocortical functioning; however, the neurophysiological and neuropsychological correlates of those differences continue to be underexplored. Informed by Evolutionary Neuroandrogenic Theory, the investigators examine the links between gender, risk-proneness, gratification delay, self-control, self-efficacy, executive functions and neurophysiological-neuroanatomical correlates in early adolescents (age 10-12 years). Participants (N=24; 50% females) will complete behavioral measurements on study constructs and perform neuropsychological tests using fMRI scanning (e.g., Go/NoGo continuous performance, stop-signal reaction time, NIH Cognition Battery, delay discounting). Female and male groups will be compared on all outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Early adolescents (age 10-12 years)
* Male and female

Exclusion Criteria:

* Gross impairment of vision or hearing that would prevent the participants from performing neuropsychological tasks
* Inability to read and follow written instructions
* WISC-V IQ score of < 80
* Physical, neurological or concurrent psychiatric impairments that could affect cognitive and motor functions
* Regular intake of medication that could alter visual, auditory, cognitive or motor functions
* History of head injury that resulted in loss of consciousness / history of brain surgery
* Current / past history of smoking and / or alcohol or drug abuse
* Absolute contraindications to undergo MRI

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Yes, participant eligibility is based on self-representation of gender identity.
Study Population: The study population will consist of healthy early adolescent (age 10-12 years) male and female subjects
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Female vs. Male differences of fMRI BOLD responses for SSRT Stop Signals | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences of functional magnetic resonance imaging reactivity of the whole brain while performing a Stop Signal Reaction Time Task
Female vs. Male differences of fMRI BOLD responses in a Go-NoGo CPT | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences of functional magnetic resonance imaging reactivity of the whole brain while performing a Go-NoGo Continuous Performance Task
Female vs. Male differences of brain structural connectivity | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences of brain structural connectivity as measured by diffusion tensor imaging and analyzed using tract-based spatial statistics
Female vs. Male differences of brain structure | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences of brain structure as determined by voxel based morphometry of structural magnetic resonance imaging data

SECONDARY OUTCOMES:
Female vs. male differences in delay discounting | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in delay discounting as measures using a delay discounting task presented on a laptop computer
Female vs. male differences in stop signal delay | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in stop signal delay of a stop signal reaction time task performed in the magnetic resonance imaging scanner
Female vs. male differences in reaction times of correct Go responses | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in reaction times of correct Go responses performed in a Go-NoGo continuous performance task performed in the magnetic resonance imaging scanner
Female vs. male differences in commission errors in a Go-NoGo CPT | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences commission errors in a Go-NoGo continuous performance task performed in the magnetic resonance imaging scanner
Female vs. male differences in Flanker Inhibitory Control and Attention Test | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in Flanker Inhibitory Control and Attention Test of the NIH Toolbox Cognition Battery
Female vs. male differences in Dimensional Change Card Sort Test | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in Dimensional Change Card Sort Test of the NIH Toolbox Cognition Battery
Female vs. male differences in Pattern Comparison Processing Speed Test | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in Pattern Comparison Processing Speed Test of the NIH Toolbox Cognition Battery
Female vs. male differences in risk-proneness | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in risk-proneness as measured by Impulsive Sensation Seeking Scale adapted by Raffaelli and Crocket (2003)
Female vs. male differences in sensation seeking | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in Brief Sensation Seeking Scale (BSSS) developed by Hoyle et al (2002)
Female vs. male differences in gratification delay | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in abbreviated 10 item Delayed Gratification Inventory (DGI-10) by Romer, Duckworth, Sznitman, & Park (2010)
Female vs. male differences in self-control | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in Perrone, Sullivan, Pratt, & Margaryan (2004) measure of self -control adapted from the Longitudinal Study of Adolescent and Adult Health (ADD Health)
Female vs. male differences in self-efficacy | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in General Self-Efficacy Scale (GSE) developed by Schwarzer & Jerusalem (1995)

OTHER OUTCOMES:
Female vs. male differences in commission errors in an SSRT | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in commission errors in a stop signal reaction time task performed in the magnetic resonance imaging scanner
Female vs. male differences in omission errors in an SSRT | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in omission errors in a stop signal reaction time task performed in the magnetic resonance imaging scanner
Female vs. male differences in omission errors in a Go-NoGo CPT | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences omission errors in a Go-NoGo continuous performance task performed in the magnetic resonance imaging scanner
Female vs. male differences in Picture Sequence Memory Test | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in Picture Sequence Memory Test of the NIH Toolbox Cognition Battery
Female vs. male differences in List Sorting Working Memory Test | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in List Sorting Working Memory Test of the NIH Toolbox Cognition Battery
Female vs. male differences in simple visual reaction time | Outcome will be measured on the first study visit (day 1) of each subject. This will also be the only time point of measurement. Outcomes of all recruited subjects within the specified study period will be considered when reporting the outcome measure.
  Female vs. male differences in a simple visual reaction time task programmed and presented in PsychoPy software environment on a laptop computer

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Trejos-Castillo, PhD, Principal Investigator — Texas Tech University; Chanaka Kahathuduwa, Study Director — Texas Tech University
Locations (1):
- Texas Tech University - Department of Human Development and Family Studies, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided